CLINICAL TRIAL: NCT01230008
Title: Adjuvant Radiotherapy in Primary Mediastinal Lymphoma in Patients That Received R-CHOP
Brief Title: Radiotherapy in Primary Mediastinal Lymphoma
Acronym: pml
Status: Completed | Type: Observational
Sponsor: Instituto Mexicano del Seguro Social (Other Government)
Responsible Party: Agustin Aviles, Mexican Institute of Social Security
Other Study IDs: katty7; katt7 (Other: Mexican Institute of Social Security)
Record Dates: First submitted 2010-10-27; First posted 2010-10-28 (Estimated); Last update posted 2010-10-28 (Estimated); Status verified 2009-06

CONDITIONS: Adjuvant Radiotherapy on Complete Remission Patients
Keywords: primary mediastinal lymphoma; radiotherapy; chemotherapy; rituximab

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Radiotherapy in mediastinal lymphoma: Adjuvant radiotherapy or not (control group) in patients treated with R-CHOP
- Radiotherapy in mediastinal lymphoma: Radiotherapy will no be administered in patients treated with R-CHOP
- Radiotherapy in primary mediastinal lymphoma: Patients with primary mediastinal lymphoma will be treated with R-CHOP as induction therapy, if complete response is achieved, they were allocated to received or no (control group) adjuvatn radiotherapy, 3.5 G to mediastinal site.
  Interventions: Radiation: no drugs

INTERVENTIONS:
Radiation: no drugs — Adjuvant radiotherapy 3.5 G will be administered or not (control group) in patients with mediastinal lymphoma,treated with R-CHOP
  Other Names: no applicable
  Groups: Radiotherapy in primary mediastinal lymphoma

SUMMARY:
The use of Rituximab has been proposed to be useful and avoid the use of radiotherapy in diffuse large B-cell lymphoma with bulky disease.We assess efficacy of adjuvant radiotherapy in patients treated with R-CHOP

ELIGIBILITY:
Inclusion Criteria:

Diagnosis of primary mediastinal lymphoma No previous treatment performance status < 2 HIV, Hepatis B and C negative Normal :Renal, hepatic, pulmonary and cardiac function

Exclusion Criteria:

pregnancy

-

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with primary mediastinal lymphoma treated in an tertiary medical center
Sampling Method: Probability Sample
Enrollment: 198 (Actual)
Dates: Start 2002-06; Primary Completion 2007-06 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
measurement of progression free-survival and overall survival at > 5 years | 5 years
  Assess if the use of adjuvant radiotherapy improve outcome in patients with primary mediastinal lymphoma treated initially with R-CHOP

SECONDARY OUTCOMES:
assess toxicity secondary to mediastinal radiotherapy | > 5 years
  Assess if the addition of mediastinal radiotherapy to patients who received anthracyclines can produce an increase in cardiac toxicity

CONTACTS AND LOCATIONS:
Locations (1):
- Oncology Research Unit, Mèxico DF, Mexico City, Mexico